CLINICAL TRIAL: NCT06440382
Title: Scottish Cervical Screening and Ethnicity Project
Acronym: SCREEN
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC19033
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2020-02

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- screening invitees: eligible women in Scotland invited to cervical screening
- interview study: 50 women from diverse ethnic groups

SUMMARY:
To identify important ethnic inequalities in cervical cancer screening participation in Scotland, and explore possible reasons for these.

DETAILED DESCRIPTION:
The 2011 Census database was linked, via the Community Health Index number, with the Scottish Cervical Screening Programme data to generate anonymised individual level information on cervical screening participation rates by self-reported ethnic group in Scotland. The cohort comprised women (aged 20 to 70) who were living in Scotland in April 2011 and took part in the 2011 Scottish census, and who were invited to participate in the Scottish Cervical Screening Programme between January 2012 and December 2018. All ethnic groups were compared to the population of White Scottish women. Qualitative interviews were carried out with 50 women (South Asian, East European, Chinese, Black African / Caribbean, or White Scottish).

ELIGIBILITY:
Inclusion Criteria:

* screening invitees through national programme

Exclusion Criteria:

* not invited to cervical screening

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women (aged 20 to 70) who were living in Scotland in April 2011 and took part in the 2011 Scottish census, and who were invited to participate in the Scottish Cervical Screening Programme between January 2012 and December 2018
Sampling Method: Probability Sample
Enrollment: 600000 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
% women who attend cervical screening | within 6 months of date of invitation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No